CLINICAL TRIAL: NCT06564818
Title: A Phase III, Placebo-Controlled, Randomized, Double-Blind Trial of Oral Doses of CYB003 to Assess Combined Safety and Efficacy in Humans With Major Depressive Disorder
Brief Title: "A Study of a Deuterated Psilocin Analog (CYB003) in Humans With Major Depressive Disorder"
Acronym: APPROACH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cybin IRL Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CYB003-002
Record Dates: First submitted 2024-08-20; First posted 2024-08-21 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-11

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; MDD; Psilocybin; Psychedelic; Psilocin; CYB003; CYB003-001; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Arm A: CYB003 in 2 of 2 Dosing Sessions (Experimental): Arm A participants will receive 16 mg of CYB003 in 2 of 2 medicine sessions, approximately three weeks apart. All Arm A participants will continue on their current antidepressants and receive psychological support throughout the study.
  Interventions: Drug: CYB003; Behavioral: Psychological Support
- Placebo Comparator Arm B: Placebo in 2 of 2 Dosing Sessions (Placebo Comparator): Arm B participants will receive placebo in 2 of 2 Dosing Sessions, approximately three weeks apart. All Arm B participants will continue on their current antidepressants and receive psychological support throughout the study. Non-responders will be eligible to receive CYB003 in a subsequent extension trial.
  Interventions: Behavioral: Psychological Support; Drug: Placebo

INTERVENTIONS:
Drug: CYB003 — CYB003 is a Deuterated Psilocin Analog.
  Arms: Experimental Arm A: CYB003 in 2 of 2 Dosing Sessions
Behavioral: Psychological Support — Manualized psychological support performed by facilitators
Drug: Placebo — Placebo
  Arms: Placebo Comparator Arm B: Placebo in 2 of 2 Dosing Sessions

SUMMARY:
The purpose of this study is to examine the efficacy, safety, and tolerability of CYB003 compared to matching placebo as adjunctive treatment in participants with MDD.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the following criteria to be included in the trial:

* Aged 18 to 85 years inclusive, at Screening
* Participant has a diagnosis of MDD (single or recurrent episode as defined by DSM-5 TR [if single episode, duration of ≥4 weeks and ≤24 months] and established as per evaluation by the Investigator. The first MDD episode must have occurred prior to age 60.
* Depression is of moderate to severe degree at Screening, independently confirmed by additional clinical assessments
* Participant has been on a stable dose of a single antidepressant medication at an adequate dose (label specified) for an adequate duration in the last 4 weeks prior to Screening and has had an inadequate response (less than 50% improvement), as judged by the Investigator and clinical interviews.
* Participant has a body mass index (BMI) of 40 kg/m2 or less (BMI ≤ 40 kg/m2), inclusive, at Screening.
* Participant is able to refrain from nicotine use during the dosing session (up to 8 hours)
* Registered with a healthcare professional who can confirm the diagnosis and previous treatments received by the participant.
* Participants capable of producing sperm must use a condom during the trial and for 12 weeks after their final dose of trial medication, if their partner is a person of childbearing potential. In addition, their partner of childbearing potential must use a highly effective method of contraception (i.e., failure rate less than 1% when used consistently and correctly) from first dosing until 12 weeks following final dosing.
* Participants of childbearing potential who have a partner capable of producing sperm must agree to use a highly effective method of contraception (i.e., failure rate less than 1% when used consistently and correctly) in combination with the use of a condom plus spermicide during the trial and for 12 weeks after their final dose of trial medication. Such participants must have a negative pregnancy test at Screening and Day -1 prior to dosing.
* Female participants who were capable of producing eggs (ova) must be postmenopausal or permanently sterile following hysterectomy, bilateral salpingectomy, and bilateral oophorectomy. Postmenopausal is defined as spontaneous amenorrhea for at least 12 months, and a serum follicle-stimulating hormone level in the menopausal range, unless the participant is taking hormone replacement therapy or is using hormonal contraception.
* Participant has provided written informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form.

Exclusion Criteria:

Participants with any of the following characteristics/conditions will be excluded from trial participation:

* Current or previously diagnosed schizophrenia spectrum or other psychotic disorders, including schizophrenia, schizoaffective disorder, schizotypal disorder, schizophreniform disorder, brief psychotic disorder, attention deficit hyperactivity disorder, current or previous history of bipolar disorder, or current borderline personality disorder.
* Family history of schizophrenia, schizoaffective disorder, or bipolar disorder type 1 (first degree relatives).
* Significant suicide risk within the past 6 months, during the Screening Period, or at Baseline; or (b) suicidal behaviors within 12 months of Screening; or (c) clinical assessment of significant suicidal risk during clinical interview; or (d) non-suicidal self-injury within 12 months of Screening.
* Current or previous diagnosis of treatment-resistant MDD, defined as failure to respond to 2 or more antidepressant treatments of 2 different classes given at an adequate dose for an adequate duration as judged by the Investigator and clinical interview.
* Has had electroconvulsive treatment, transcranial magnetic stimulation, deep brain stimulation, or vagal nerve stimulation for any episode of MDD in the last 6 months.
* Currently receiving a monoamine oxidase inhibitor, tricyclic antidepressant, mirtazapine, trazodone, moclobemide, buspirone, ketamine or S-ketamine, or an antipsychotic or mood stabilizer for MDD.
* Participant report of (or if available in medical record) exposure to psilocin, or 5-HT2a receptor agonists, or any other psychedelics, such as ayahuasca, mescaline, lysergic acid diethylamide, peyote, or 3,4-methylenedioxymethamphetamine, more than 4 times over the participant's lifetime or any psychedelic use within 12 months prior to Screening.
* Clinically relevant history of abnormal physical health interfering with the trial as determined by medical history and physical examinations obtained during Screening as judged by the Investigator (including but not limited to, neurological, cardiovascular, respiratory, gastrointestinal [including dyspepsia or gastroesophageal reflux disease], hepatic, or renal disorder).
* Participants with renal insufficiency.
* Has hypothyroidism or hyperthyroidism, unless controlled on appropriate medication with no change in dosage for at least 12 weeks prior to Screening.
* Current diagnosis of uncontrolled hypertension or an arrhythmia, or clinically relevant abnormal results for heart rate or blood pressure
* History or clinical evidence of any disease and/or existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism, or excretion of the trial medication.
* Participant has a presence or relevant history of organic brain disorders (e.g., epilepsy, seizure, intracranial hypertension, intracranial bleed and aneurysmal disease, brain tumor or other medical conditions associated with seizures or convulsions).
* Known sensitivity to psilocin and/or any excipients present in the formulation.
* Participant is taking or has taken OTC doses of 5 hydroxytryptophan or St John's Wort within 45 days prior to trial medication administration.
* Strenuous exercise within 48 hours prior to each clinic visit.
* The participant has participated in a clinical trial and has received a medication or a new chemical entity within 12 weeks prior to dosing of current trial medication.
* Participants capable of producing sperm who will not abstain from sperm donation between first dosing and 12 weeks after final dosing.
* Participants of childbearing potential who are pregnant, breastfeeding, planning to conceive or unwilling to abstain from egg (ova) donation between first dosing and 12 weeks after final dosing.
* History of serotonin syndrome.
* Unwilling to consent to audio and video recording of psychological support and dosing sessions.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | Screening Day-45, Baseline Day-1, Day 2, Day 10, Day 21, Day 23, Day 31, and Day 42 (End of Treatment)
  The MADRS is a 10-item scale with ratings based on a clinical interview which moves from broadly phrased questions about symptoms to more detailed ones allowing a precise rating of severity.

SECONDARY OUTCOMES:
The Beck Depression Inventory-Second Edition (BDI-II) | Baseline Day-1, Day 21, and Day 42 (End of Treatment)
  The Beck Depression Inventory-Second Edition (BDI-II) is a 21-question multiple-choice self-report inventory, assessing depressive symptoms and severity.
The Clinical Global Impression Scale (CGI-S) | Screening Day-45, Baseline Day-1, and Day 42 (End of Treatment)
  The Clinical Global Impression Scale is a clinician-rated instrument comprised of 3 global measures: severity of illness, global improvement, and efficacy index. Only the severity of illness and global improvement measures will be utilized for this trial.
The Generalized Anxiety Disorder 7-item scale (GAD-7) | Baseline Day-1, Day 21, and Day 42 (End of Treatment)
  The Generalized Anxiety Disorder 7-item scale (GAD-7) is a 7-item self-reported assessment that measures the severity of generalized anxiety disorder symptoms.
The Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) | Baseline Day-1, Day 21, and Day 42 (End of Treatment)
  The original Quality of Life Enjoyment and Satisfaction Questionnaire is a 93 item, participant facing, self-reported measure used to evaluate intervention-related changes in quality of life, divided into the following sections: physical health, feelings, work, household duties, school, leisure time activities, social relations, and general activities. The Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) version will be used in this trial.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Chair — Cybin IRL Limited
Locations (45):
- United States (45):
  - Scottsdale Research Institute, Phoenix, Arizona
  - Mountain Clinical Trials, Phoenix, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Del Sol Research Management, Tucson, Arizona
  - CenExel CIT (Clinical Innovations, Inc), Bellflower, California
  - Kadima Neuropsychiatry Institute, La Jolla, California
  - Bespoke Treatment/Lipov Medical Group, Los Angeles, California
  - Catalina Research Institute, Montclair, California
  - Excell Research, Inc, Oceanside, California
  - Open Mind Collective/UCSF Medical Center Mount Zion, San Francisco, California
  - Inland Psychiatric Medical Group Inc, San Juan Capistrano, California
  - Mountain View Clinical Research, Denver, Colorado
  - Starlight Clinical Research, Evergreen, Colorado
  - Research Centers of America, Hollywood, Florida
  - K2 Medical Research-Maitland, Maitland, Florida
  - Floridian Neuroscience Institute, Miami, Florida
  - Innovative Clinical Research, INC, North Miami, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Charter Research, Orlando, Florida
  - Combined Research Orlando Phase I-IV, Orlando, Florida
  - K2 Medical Research - Tampa, Tampa, Florida
  - Atlanta Center for Medical Research, CenExel, Atlanta, Georgia
  - CenExel iResearch Atlanta, Decatur, Georgia
  - CenExel iResearch Savannah, Savannah, Georgia
  - Great Lakes Clinical Trials, DBA Flourish Research, Chicago, Illinois
  - Uptown Research Institute, Chicago, Illinois
  - Psychiatric Medicine Associates, LLC, Skokie, Illinois
  - DelRicht Research, New Orleans, Louisiana
  - Sunstone Medical, PC, Rockville, Maryland
  - Adams Clinical Boston, Boston, Massachusetts
  - Adams Clinical, Boston, Massachusetts
  - Elixia Health, Springfield, Massachusetts
  - Redbird Research, LLC, Las Vegas, Nevada
  - Oasis Clinical Trials, Las Vegas, Nevada
  - Global Medical Institutes, Princeton Medical Institute, Princeton, New Jersey
  - Adams Clinical Harlem, New York, New York
  - Adams Clinical Bronx, The Bronx, New York
  - Monroe Biomedical Research, Monroe, North Carolina
  - Neurobehavioral Clinical Research, North Canton, Ohio
  - Clinical Neuroscience Solutions, CNS Healthcare, Memphis, Tennessee
  - InSite Clinical Research, LLC, DeSota, Texas
  - Zillan Clinical Research, Houston, Texas
  - AIM Trials, Plano, Texas
  - Cedar Clinical Research, Murray, Utah
  - Inner Space Research, LLC, Orem, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Apply for Trial Here — https://www.approach-mdd-trial.com/